CLINICAL TRIAL: NCT03024411
Title: Music and/or Video Games for Pain Management During Induction of Labor
Brief Title: Music and/or Video Games During Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-0071
Record Dates: First submitted 2016-03-14; First posted 2017-01-18 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music/video games (Experimental): iPod (Music/video games)
  Interventions: Other: iPod (Music/video games)
- No intervention (No Intervention): No intervention

INTERVENTIONS:
Other: iPod (Music/video games) — Experimental patients will be given an iPod to enjoy music/video games during induction of labor.
  Arms: Music/video games

SUMMARY:
Data are lacking regarding the use of music and video games for the management of pain in labor. Pregnant women that are scheduled for labor induction with Foley bulb after 37 weeks will be approached for participation in the study. Patients will be randomized to a music/video games group and a non-music/video games group. Those randomized to group with music/video games will be given an iPod for those purposes.The primary outcome will be the time for patients to request pain medications after Foley bulb placement. The two groups will be compared for differences in pain outcomes.

DETAILED DESCRIPTION:
For decades, investigators have been evaluating the efficacy of music for pain relief. Music for pain management has been studied in the field of palliative care, oncology, physical therapy, pediatrics, post-operative procedural pain and childbirth. A 2006 Cochrane review found that listening to music reduces pain intensity levels and opioid requirements, but the magnitude of the benefits is small and the clinical importance unclear. Previous studies in obstetrics vary, as some evaluate music for pain control at time of cesarean section and others during labor. A 2014 study investigated the effect of progressive muscle relaxation exercises and music on low back pain and quality of life in pregnancy. Some previous studies investigating music or white noise for pain control during labor revealed beneficial results. One prospective trial of 25 women found little practical value of audio-analgesia.

However, most studies evaluating music therapy for pain relief in labor were limited by sample size. Specifically, a 2011 Cochrane review investigating randomized controlled trials comparing relaxation methods as a method of pain management in labor found insufficient evidence for the role of music and audio-analgesia and the need for further research. Excluded from this review was a trial by Phumdoung et al. due to the inability to obtain additional methodological and statistical information from the authors. More recently, a randomized controlled trial (RCT) done in Turkey randomized 156 women into a music and control group. Mothers in the music group were found to have a significantly lower level of pain and anxiety in all stages of labor. Pain and anxiety were evaluated by a visual analog scale. While this evidence is the best to date, there is a lack of generalizability for other populations and the primary outcome was subjective. A 2012 systematic review of video games found improvement in psychological therapy, physical therapy, physical activity, clinical skills, health education, pain distraction, and disease self-management outcomes.

Labor induction is a common obstetrical procedure. Labor results in severe pain for many women and typically requires medical treatment for pain relief. Types of analgesia for pain control on labor include parenteral (Fentanyl, Nalbuphine, Meperidine) and regional (spinal, epidural, combined spinal epidural) analgesia. However, all types of analgesia pose risks to the mother and fetus. Administration of parenteral agents result in minimal-to-absent reduction in pain scores and high doses affect fetal heart rate tracing and later increase the number of infants requiring naloxone therapy. While regional analgesia provides superior pain relief, common complications include hypotension, fever, postdural puncture headache, transient fetal heart rate decelerations, pruritus, and inadequate pain relief. Due to these risks and other reasons, many women prefer to go through labor without medical therapies or with minimal medical therapy and desire complementary therapies to help manage their pain. Data are lacking regarding the use of music and video games for the management of pain in labor.

In view of the lack of good quality evidence from well designed RCTs, we propose a randomized controlled trial to determine the utility of music and video games for pain management during induction of labor. Pregnant women that are scheduled for labor induction with Foley bulb after 37 weeks will be approached for participation in the study. The study informed consent will be obtained. Patients will be randomized to a music/video games group (group 1) and a non-music/video games group (group 2). Those randomized to group with music/video games will be given an iPod for those purposes. The iPod will include free music applications such as Pandora as well as some of the most commonly downloaded games. Randomization will be performed using a computer generated random list of numbers assigning patients to the 2 groups of the study. Randomization will occur after the Foley bulb is placed. Study assignment and the list of random number assignments will be kept secure in opaque envelopes until the end of the study.

Prospective subjects presenting for induction of labor in labor and delivery, and willing to participate in the study will be evaluated for their eligibility. After the Foley bulb is placed, patients will be randomized. Those assigned to the music/video game group will be given an iPod to use during labor. These patients will have the choice of listening to music via earphones or a speaker which amplifies the sound. Patients assigned to the non-music/video game group will not be given an iPod and will be asked to avoid using their own personal devices (if applicable) as much as possible. Understanding that patients randomized to the non-music/video game may still elect to use their own electronic devices, time of use of electronics for music/video game purposes will be recorded in both groups with assistance from the patients and nursing staff.

All nurses will be educated regarding the study procedure. Nurses will not ask any patient if they desire pain medicine to avoid prompting the patient. Every patient enrolled will receive a Foley bulb inserted just superior to the internal cervical os and then inflated with normal saline for mechanical dilation of the cervix. The Foley bulb will be placed under traction by taping the tubing to the patient's leg. No additional traction will be applied to the Foley bulb after placement and initial traction. After twelve hours, if the Foley balloon is still in place, the Foley balloon will be deflated and removed and the remainder of obstetrical care will be left to the discretion of the supervising faculty. After six hours or after epidural placement the use of music/video games will be continued or ceased pending patient desire.

The study will be explained as in the consent form and if agreed, patients will elect either to participate in the study or not after all risks and benefits are explained. Data to be collected will consist of age, gravida/para, gestational age, body mass index, time and date of intervention, time and date of delivery, mode of delivery, bishop score at admission (bishop score is a score that assesses cervical readiness for delivery and is measured by digital pelvic exam. A score < 7 is considered unfavorable and is an indication for cervical ripening to induce labor), time and date of pain medication request, type and amount of parenteral medication, time from Foley bulb placement until expulsion, patient pain score by visual analog scale, and patient satisfaction. Data will be extracted from patients' medical records as well as from direct interview with the patient. If elected to participate consents will be obtained and stored in patient chart. A copy of the consent will be given to the patient. Patients will be consented in either English or Spanish by research personnel fluent in the language. The primary outcome will be the time for patients to request pain medications after Foley bulb placement. The two groups will be compared for differences in pain outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years old
* Pregnant women > or = 37 weeks gestation
* Induction of labor using Foley bulb
* Singleton gestation
* Vertex fetal presentation
* Intact membranes

Exclusion Criteria:

* Any contraindication for vaginal delivery (malpresentation, placenta previa)
* Previous cesarean section
* Gestational age <37 weeks gestation
* Receiving pain medication at time of Foley bulb placement
* Chronic narcotic use (methadone, suboxone, oxycodone, etc.)
* Visual or auditory impairment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2017-07-08 (Actual); Study Completion 2017-08-04 (Actual)

PRIMARY OUTCOMES:
Time until patient request for pain medication after Foley bulb placement. | From time of Foley bulb placement (randomization) until time of request for pain medicine or time of delivery, whichever came first, assessed up to 3 days.
  Time from Foley bulb placement until patient requests pain medication.

SECONDARY OUTCOMES:
Parenteral medication | From time of Foley bulb placement (randomization) until time of delivery, assessed up to 3 days.
  Amount of parenteral medication administered
Visual analog scale (VAS) pain score | Six hours from time of Foley bulb placement (randomization).
  Visual analog scale (VAS) pain score every hour for the first 6 hours after Foley bulb placement.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Dixon, M.D., Principal Investigator — The University of Texas Medical Branch at Galveston
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Background] Smith CA, Levett KM, Collins CT, Crowther CA. Relaxation techniques for pain management in labour. Cochrane Database Syst Rev. 2011 Dec 7;(12):CD009514. doi: 10.1002/14651858.CD009514. PMID 22161453
- [Background] van der Heijden MJ, Oliai Araghi S, van Dijk M, Jeekel J, Hunink MG. The Effects of Perioperative Music Interventions in Pediatric Surgery: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. PLoS One. 2015 Aug 6;10(8):e0133608. doi: 10.1371/journal.pone.0133608. eCollection 2015. PMID 26247769
- [Background] Hsieh C, Kong J, Kirsch I, Edwards RR, Jensen KB, Kaptchuk TJ, Gollub RL. Well-loved music robustly relieves pain: a randomized, controlled trial. PLoS One. 2014 Sep 11;9(9):e107390. doi: 10.1371/journal.pone.0107390. eCollection 2014. PMID 25211164
- [Background] Hartling L, Newton AS, Liang Y, Jou H, Hewson K, Klassen TP, Curtis S. Music to reduce pain and distress in the pediatric emergency department: a randomized clinical trial. JAMA Pediatr. 2013 Sep;167(9):826-35. doi: 10.1001/jamapediatrics.2013.200. PMID 23857075
- [Background] Primack BA, Carroll MV, McNamara M, Klem ML, King B, Rich M, Chan CW, Nayak S. Role of video games in improving health-related outcomes: a systematic review. Am J Prev Med. 2012 Jun;42(6):630-8. doi: 10.1016/j.amepre.2012.02.023. PMID 22608382
- [Background] MOORE WM, BROWNE JC, HILL ID. CLINICAL TRIAL OF AUDIO-ANALGESIA IN CHILDBIRTH. J Obstet Gynaecol Br Commonw. 1965 Aug;72:626-9. doi: 10.1111/j.1471-0528.1965.tb00074.x. No abstract available. PMID 14341119
- [Background] Yinger OS, Gooding LF. A systematic review of music-based interventions for procedural support. J Music Ther. 2015 Spring;52(1):1-77. doi: 10.1093/jmt/thv004. Epub 2015 Apr 15. PMID 25878063
- [Background] Cepeda MS, Carr DB, Lau J, Alvarez H. Music for pain relief. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD004843. doi: 10.1002/14651858.CD004843.pub2. PMID 16625614
- [Background] Browning CA. Using music during childbirth. Birth. 2000 Dec;27(4):272-6. doi: 10.1046/j.1523-536x.2000.00272.x. PMID 11251514
- [Background] Akmese ZB, Oran NT. Effects of Progressive Muscle Relaxation Exercises Accompanied by Music on Low Back Pain and Quality of Life During Pregnancy. J Midwifery Womens Health. 2014 Sep-Oct;59(5):503-9. doi: 10.1111/jmwh.12176. Epub 2014 Jun 25. PMID 24965313
- [Background] Wright J, Adams D, Vohra S. Complementary, holistic, and integrative medicine: music for procedural pain. Pediatr Rev. 2013 Nov;34(11):e42-6. doi: 10.1542/pir.34-11-e42. No abstract available. PMID 24187147
- [Background] Keenan A, Keithley JK. Integrative Review: Effects of Music on Cancer Pain in Adults. Oncol Nurs Forum. 2015 Nov;42(6):E368-75. doi: 10.1188/15.ONF.E368-E375. PMID 26488843
- [Background] BURT RK, KORN GW. AUDIOANALGESIA IN OBSTETRICS. "WHITE SOUND" ANALGESIA DURING LABOR. Am J Obstet Gynecol. 1964 Feb 1;88:361-6. No abstract available. PMID 14123408
- [Background] Tsai HF, Chen YR, Chung MH, Liao YM, Chi MJ, Chang CC, Chou KR. Effectiveness of music intervention in ameliorating cancer patients' anxiety, depression, pain, and fatigue: a meta-analysis. Cancer Nurs. 2014 Nov-Dec;37(6):E35-50. doi: 10.1097/NCC.0000000000000116. PMID 24662723
- [Background] Bellieni CV, Cioncoloni D, Mazzanti S, Bianchi ME, Morrone I, Becattelli R, Perrone S, Buonocore G. Music provided through a portable media player (iPod) blunts pain during physical therapy. Pain Manag Nurs. 2013 Dec;14(4):e151-e155. doi: 10.1016/j.pmn.2011.09.003. Epub 2011 Nov 16. PMID 24315267
- [Background] Gutgsell KJ, Schluchter M, Margevicius S, DeGolia PA, McLaughlin B, Harris M, Mecklenburg J, Wiencek C. Music therapy reduces pain in palliative care patients: a randomized controlled trial. J Pain Symptom Manage. 2013 May;45(5):822-31. doi: 10.1016/j.jpainsymman.2012.05.008. Epub 2012 Sep 24. PMID 23017609
- [Background] Li Y, Dong Y. Preoperative music intervention for patients undergoing cesarean delivery. Int J Gynaecol Obstet. 2012 Oct;119(1):81-3. doi: 10.1016/j.ijgo.2012.05.017. Epub 2012 Jul 15. PMID 22795881
- [Background] Phumdoung S, Good M. Music reduces sensation and distress of labor pain. Pain Manag Nurs. 2003 Jun;4(2):54-61. doi: 10.1016/s1524-9042(02)54202-8. PMID 12836149
- [Background] Liu YH, Chang MY, Chen CH. Effects of music therapy on labour pain and anxiety in Taiwanese first-time mothers. J Clin Nurs. 2010 Apr;19(7-8):1065-72. doi: 10.1111/j.1365-2702.2009.03028.x. PMID 20492051
- [Background] Simavli S, Gumus I, Kaygusuz I, Yildirim M, Usluogullari B, Kafali H. Effect of music on labor pain relief, anxiety level and postpartum analgesic requirement: a randomized controlled clinical trial. Gynecol Obstet Invest. 2014;78(4):244-50. doi: 10.1159/000365085. Epub 2014 Sep 16. PMID 25227477
- [Background] American College of Obstetrics and Gynecology. ACOG practice bulletin. Obstetric analgesia and anesthesia. Number 36, July 2002. American College of Obstetrics and Gynecology. Int J Gynaecol Obstet. 2002 Sep;78(3):321-35. doi: 10.1016/s0020-7292(02)00268-0. PMID 12452132
- [Derived] Dixon CL, Monsivais L, Chamseddine P, Olson G, Pacheco LD, Saade GR, Costantine MM. The Effect of Distraction during Labor Induction on Timing of Analgesia Request: A Randomized Clinical Trial. Am J Perinatol. 2019 Nov;36(13):1351-1356. doi: 10.1055/s-0038-1676974. Epub 2019 Jan 4. PMID 30609428